CLINICAL TRIAL: NCT05439395
Title: Multi Center, International, Single-arm, Retrospective, Observational Post Market Clinical Follow-Up (PMCF) Study on the Clinical Performance of Steelex® Sternum Set for Sternal Closure in Patients Undergoing Cardiac Surgery
Brief Title: Study on the Clinical Performance of Steelex® Sternum Set for Sternal Closure
Acronym: STERCCAS
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2028
Record Dates: First submitted 2022-06-22; First posted 2022-06-30 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Cardiac Valve Insufficiency; Aortic Valve Stenosis
Keywords: Median Sternotomy; Partial Sternotomy; Coronary Artery Bypass Grafting (CABG); Cardiac Valve Replacement; Cardiac Valve Reconstruction
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEELEX: Steelex® Sternum Set for sternal closure
  Interventions: Device: Sternum Closure after Cardiac Surgery

INTERVENTIONS:
Device: Sternum Closure after Cardiac Surgery — Sternal closure using Steelex® Sternum Set after CABG or cardiac valve replacement / reconstruction.

SUMMARY:
The study is designed as a retrospective, international, multi-center cohort study to evaluate Steelex® Sternum Set for sternum closure. The data from 2 clinics located in Germany and Spain participating in the "OPTICABG" as well as in the "PREMIVALVE" study will be used for assessment. Only patients receiving a complete or a partial sternotomy closed with Steelex® Sternum Set will be included in the analysis. "OPTICABG" patients were followed up 3 months after surgery and "PREMIVALVE" patients until 6 months after surgery. Adverse Events (AE) / Serious Adverse Events (SAE)(e.g. surgical site infection, sternum stability, stroke, myocardial infraction, death etc.) reported in both studies will be used for the STERCCAS analysis.

ELIGIBILITY:
Inclusion Criteria:

* OPTICABG study patients undergoing an elective, primary coronary artery bypass graft surgery (CABG) receiving a sternotomy, by whom the sternum was closed using Steelex® Sternum Set.
* PREMIVALVE study patients undergoing a cardiac valve replacement or reconstruction receiving a complete or partial sternotomy, by whom the sternum was closed using Steelex® Sternum Set.
* Eligible patients from the OPTICABG study and PREMIVALVE study who have provided their written informed consent
* Age ≥18 years

Exclusion Criteria:

* OPTICABG and PREMIVALVE patients receiving a sternotomy or partial sternotomy which was not closed with Steelex® Sternum Set.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a partial or a complete sternotomy closed with Steelex Sternum Set participating either in the OPTICABG or PREMIVALVE study.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Incidence of a composite endpoint consisting of sternum instability, sternum dehiscence, superficial and deep sternal wound infection | up to 6 months after surgery
  Combination of:
  * Incidence of sternum instability
  * Incidence of sternum dehiscence
  * Incidence of superficial and deep sternal wound infection according to classification of Centers for Disease Control and Prevention (CDC)

SECONDARY OUTCOMES:
Incidence of sternum instability | up to 6 months after surgery
  Number of patients presenting with instability of the sternum after sternal closure with Steelex® Sternum Set
Incidence of sternum dehiscence | up to 6 months after surgery
  Number of patients presenting with dehiscence of the sternum after sternal closure with Steelex® Sternum Set
Incidence of superficial and deep sternal wound infection | up to 6 months after surgery
  Number of patients presenting with superficial and deep sternal wound infection according to CDC classification after sternal closure with Steelex® Sternum Set
Incidence of other cardiac and cerebral complications | up to 6 months after surgery
  Number of patients presenting with other cardiac and cerebral complications such as stroke, myocardial infarction, death, as well as mediastinitis after sternal closure with Steelex® Sternum Set
Incidence of suture related complications | up to 6 months after surgery
  Number of patients presenting with suture related complications (e.g. wire breakage) after sternal closure with Steelex® Sternum Set
Length of hospital stay | until discharge (approximately 10 days postoperative)
  Number of days the patient has to stay in hospital
Length of intensive care unit stay | until discharge (approximately 10 days postoperative)
  Number of days the patient has to stay in intensive care unit after intervention
Health Status measured with EQ-5D-5L Score | up to 6 months after surgery
  EQ-5D-5L is a Quality of Life Score introduced by the EuroQol Group. The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  Descriptive system comprises five dimensions (5D): mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels (5L): no problems, slight problems, moderate problems, severe problems, extreme problems. Each answer results in a 1-digit number. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Intraoperative handling of the Steelex® Sternum Set | at time of surgery
  the handling is examined using a survey, which will be answered and filled out prospectively and anonymously once by all involved cardiac surgeons

CONTACTS AND LOCATIONS:
Locations (2):
- Robert Bosch KH Stuttgart, Stuttgart, Germany
- Hospital de la Santa Creu I Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No